CLINICAL TRIAL: NCT02640144
Title: The Influence of Hyaluronic Acid Injection Following Knee Arthroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Medical Center (Other)
Responsible Party: Principal Investigator, Noam Reshef, Attending Orthopedic Surgeon, Orthopedic Sports specialist, Ziv Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0013-15-ZIV
Record Dates: First submitted 2015-12-10; First posted 2015-12-28 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cartilage Damage
Keywords: Hyaluronic acid; Knee arthroscopy; pain reduction; swelling; osteoarthritis; cartilage lesion; rehabilitation following knee arthroscopy; Hyaluronic acid injection
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Randomized, patients that are going for knee arthroscopy for any indication including pain and cartilage damage or osteoarthritis. After surgery - will receive 3 injections of Sodium Hyaluronate 1% - ARTHREASE TM
  Interventions: Drug: Sodium Hyaluronate 1%
- Control group (Placebo Comparator): Randomized, patients that are going for knee arthroscopy for any indication including pain and cartilage damage or osteoarthritis. After surgery - will receive 3 injections of BPS - Buffer Phosphate Solution - as a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Hyaluronate 1% — Intra articular knee injection following arthroscopy
  Other Names: ARTHREASE; Euflexxa
  Arms: Treatment group
Drug: Placebo — Intra articular knee injection following knee arthroscopy. Serves as a placebo. This is the actual buffer of the ARTHREASE injection.
  Other Names: BPS = Buffer Phosphate Solution
  Arms: Control group

SUMMARY:
This is a prospective, double blind randomized controlled trial. In this study we will investigate the influence of hyaluronic acid injection to knee after knee arthroscopy, when known or discovered cartilage damage greater than International Cartilage Research Society score (ICRS) grade 2 is found. The indication for arthroscopy is not necessarily the cartilage damage. A set of 3 consecutive injections will be administered and follow up of physical examination and questionaries will be done.

Our null hypothesis is that the administration of hyaluronic acid will show decrease pain and quicker rehabilitation and return to normal activity in patients with grade 2 and higher cartilage damage that had gone through knee arthroscopy.

DETAILED DESCRIPTION:
The use of hyaluronic acid is well known as one of the treatment modalities for knee osteoarthritis (OA) .Arthroscopy is a controversial treatment option for knee OA but in some cases, during knee arthroscopy done for other indication, cartilage damage is noted. This cartilage damage may slower the healing and rehabilitation process after knee arthroscopy. Therefore we will evaluate the influence of hyaluronic acid injection on the healing and rehabilitation process following knee arthroscopy.

All patients will be recruited prior to the arthroscopy. All patients will sign a concent form.Patients will be randomly divided to 2 groups which are the 2 arms of this study - treatment group and control group. All patient will be examined by a senior orthopedic surgeon and will fill the pre operative questionnaires. MRI scan of the operated knee prior for the surgery will be collected and evaluated.Knee arthroscopy will be performed by 2 senior orthopedic surgeons. Data and arthroscopic findings will be collected and documented during surgery. 2 weeks after surgery patients will be evaluated in the hospitals' outpatients clinic. The treatment group will be given a series of 3 injections of Sodium Hyaluronate 1%(ARTHREASE, TM) - one injection per week. The control group will be given a series of 3 injections of placebo (BPS - Buffer Phosphate Solution - the buffer solution of the hyaluronic acid regular injections). The syringes will be blinded to the patients and the physician.

questionnaires will be given at 2 weeks, 6 weeks, 3months and 6 months post operatively

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* signing a concent form
* Assigned for knee arthroscopy.
* Known chondral lesion of at least ICRS grade 2 in one or mor of the knee compartments per MRI prior to knee arthroscopy.
* Cartilage lesion of at least ICRS grade 2 in one or mor of the knee compartments that was found during the knee arthroscopy.

Exclusion Criteria:

* Rheumatic disease
* Synovial disease such as (but not limited to) Pigmented ViloNodular synovitis (PVNS)
* Infection of the operated knee - new or previous
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | up to 6 month
  The treatment group will show lower scores than control group at all checkpoints- 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Evaluated using Visual Analog Scale (VAS) for pain
Change in the International Knee Documentation Committee (IKDC) score as a measure of Return to normal activity | up to 6 month
  The treatment group will show quicker return to normal activity that control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Evaluation is using the International Knee Documentation Committee (IKDC) score
Change in the knee circumference as a measure for Knee swelling | up to 6 month
  The treatment group will show less episodes of knee swelling than the control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Will be evaluated by measuring the knee circumference using a simple measuring tape in centimeters.
Change in "Tegner-Lysholm" score as a measure of better function | up to 6 month
  The treatment group will show better scores in all functional questionnaires than the control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively.The questionnaires that will be used is "Tegner - Lysholm" score
Change in the Short Form (SF) 12 score as a measure of return to normal activity | up to 6 months
  The treatment group will show quicker return to normal activity that control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Evaluation is using Short Form (SF)-12 score.
Subjective description of return to normal activity as described by patients | up to 6 months
  The treatment group will show quicker return to normal activity that control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Evaluation is subjective by patients description.
Change in the "Tegner-Lysholm" score as a measure of return to normal activity | up to 6 months
  The treatment group will show quicker return to normal activity that control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Evaluation is subjective by using "Tegner - Lysholm" score
Subjective change in knee swelling | up to 6 months
  The treatment group will show less episodes of knee swelling than the control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively. Will be evaluated subjectively by the patients description.
Change in Short Form(SF) 12 score as a measure of better function | up to 6 months
  The treatment group will show better scores in all functional questionnaires than the control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively.The questionnaires that will be used is Short-Form (SF)12 score
Change in the International Knee Documentation Committee (IKDC) score as a measure of better function | up to 6 months
  The treatment group will show better scores in all functional questionnaires than the control group at all checkpoints - 2 weeks post operatively, 6 weeks post operatively, 3 months post operatively and 6 months post operatively.The questionnaires that will be used is International Knee Documentation Committee (IKDC) score

CONTACTS AND LOCATIONS:
Overall Officials: Noam Reshef, MD, Principal Investigator — Ziv Medical Center, Zefat, Israel

REFERENCES:
- [Background] Leighton R, Akermark C, Therrien R, Richardson JB, Andersson M, Todman MG, Arden NK; DUROLANE Study Group. NASHA hyaluronic acid vs. methylprednisolone for knee osteoarthritis: a prospective, multi-centre, randomized, non-inferiority trial. Osteoarthritis Cartilage. 2014 Jan;22(1):17-25. doi: 10.1016/j.joca.2013.10.009. Epub 2013 Nov 1. PMID 24185114
- [Background] Witteveen AG, Sierevelt IN, Blankevoort L, Kerkhoffs GM, van Dijk CN. Intra-articular sodium hyaluronate injections in the osteoarthritic ankle joint: effects, safety and dose dependency. Foot Ankle Surg. 2010 Dec;16(4):159-63. doi: 10.1016/j.fas.2009.10.003. Epub 2009 Nov 8. PMID 21047602
- [Background] Kirchner M, Marshall D. A double-blind randomized controlled trial comparing alternate forms of high molecular weight hyaluronan for the treatment of osteoarthritis of the knee. Osteoarthritis Cartilage. 2006 Feb;14(2):154-62. doi: 10.1016/j.joca.2005.09.003. Epub 2005 Oct 19. PMID 16242361
- [Result] Thein R, Haviv B, Kidron A, Bronak S. Intra-articular injection of hyaluronic acid following arthroscopic partial meniscectomy of the knee. Orthopedics. 2010 Oct 11;33(10):724. doi: 10.3928/01477447-20100826-11. PMID 20954664
- [Result] Altman RD, Rosen JE, Bloch DA, Hatoum HT, Korner P. A double-blind, randomized, saline-controlled study of the efficacy and safety of EUFLEXXA for treatment of painful osteoarthritis of the knee, with an open-label safety extension (the FLEXX trial). Semin Arthritis Rheum. 2009 Aug;39(1):1-9. doi: 10.1016/j.semarthrit.2009.04.001. Epub 2009 Jun 17. PMID 19539353
- Available data/document: Study Protocol — http://www.nr-ortho.com — Original study protocol is written in Hebrew. protocol is available at the Ziv Medical Center, Institutional Review Board (IRB) , or in direct request via the website address posted above.